CLINICAL TRIAL: NCT01188408
Title: A Multicenter, Open-Label, Phase II Study of LE-DT for Efficacy and Safety in Patients With Metastatic Castrate Resistant Prostate Cancer
Brief Title: Efficacy and Safety Study of LE-DT to Treat Metastatic Castrate Resistant Prostate Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study shut-down in 12/2010 when NeoPharm merged with Insys.
Sponsor: INSYS Therapeutics Inc (Industry)
Responsible Party: Aquilur Rahman, NeoPhram, Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LE-DT 201
Record Dates: First submitted 2010-08-19; First posted 2010-08-25 (Estimated); Last update posted 2018-03-12 (Actual); Status verified 2018-03

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Liposome Entrapped Docetaxel (LE-DT) (Experimental): Disease status and tumor responses/progression is assessed in accordance to the RECIST guideline
  Interventions: Drug: Liposome Entrapped Docetaxel (LE-DT)

INTERVENTIONS:
Drug: Liposome Entrapped Docetaxel (LE-DT) — 110 mg/m2 IV (in vein) on day 1 of each 21 day cycle, 6 cycles or until disease progression or unacceptable toxicity
  Other Names: LE-DT; Liposomal Docetaxel

SUMMARY:
LE-DT is a novel, proprietary delivery system of docetaxel developed by NeoPharm, Inc. Docetaxel (currently marketed as Taxotere) is an anti-microtubular network agent and is one of the most active agents in the treatment of metastatic castrate resistant prostate cancer (CRPC) and other variety of cancers. Taxotere has poor solubility and is designed to be administered with Tween 80 in ethanol. This vehicle causes acute hypersensitivity reaction. By removing toxic detergent used in Taxotere, the form of LE-DT, shows reduced toxicity and comparable therapeutic efficacy in pre-clinical study. The clinical evidence obtained from the NeoPharm Phase I study shows fewer side effects and possibly administered at higher dose to induce greater effectiveness of LE-DT. The current Phase II study is designed to accomplish the following objectives:

1. Assess the antitumor effect indicator serum prostate specific antigen (PSA) following the intravenous (IV) administration of 110 mg/m2 LE-DT every three weeks in patients with metastatic castrate resistant prostate cancer
2. To evaluate the measurable soft tissue disease response using the response evaluation criteria in solid tumor (RECIST) methodology
3. To evaluate the progression-free survival (PFS) and overall survival (OS)
4. To correlate PSA expression with tumor response
5. To evaluate the safety of LE-DT at 110 mg/m2 level, in particular peripheral neuropathy, water retention as well as myelotoxicity
6. To evaluate the quality of life (QOL)

ELIGIBILITY:
Inclusion Criteria:

1. Be 18 years or older and male.
2. Have histologically or cytologically confirmed diagnosis of adenocarcinoma of the prostate.
3. Patients without evidence of PSA progression must have clinical or radiographic evidence of metastatic disease.
4. Must have castrate levels of testosterone (serum testosterone less than 50ng/dl) by either being on androgen ablation therapy with a luteinizing hormone-releasing hormone (LHRH) agonist or have had a prior bilateral orchiectomy.
5. Patients must have documented evidence of disease progression: progressive disease is defined as a minimum of three consecutive elevations in PSA each obtained a minimum of one week apart with the last value being greater than 2 ng/mL and/or new metastatic lesions on bone scan (minimum of 2) and/or new or progressive disease on CT or MRI scan.
6. For patients on an antiandrogen (flutamide, nilutamide, bicalutamide)

   1. If given as part of first line therapy or for patients who did respond to antiandrogen second line therapy, the patient must demonstrate progression of disease at least 4 weeks beyond discontinuation of such agents to rule out an antiandrogen withdrawal response.
   2. If given as a second line therapy and the patient did not respond or had a decline in PSA for less than 3 months, it is not required to observe for a withdrawal response.
7. Chemotherapy-naïve patients (unlimited prior regimens of hormonal therapy are acceptable).
8. Have no other malignancy within the past five years, except non-melanoma, skin cancer.
9. Have recovered from acute toxicities of prior treatment:

   1. Greater than or equal to 4 weeks must have elapsed since receiving hormonal therapy (except for chronic non-investigational gonadotropin releasing hormone analogs or other primary androgen suppressive therapy which are required), biologic agents or any investigational agent (palliative bisphosphonate therapy for bone pain can be administered as clinically indicated).
   2. Greater than or equal to 4 weeks must have elapsed since receiving any radiotherapy
   3. Greater than or equal to 2 weeks must have elapsed since any prior surgery or granulocyte-stimulating growth factor therapy.
10. Have the following hematology levels at Baseline:

    1. Absolute Neutrophil Count (ANC) greater than or equal to1,500 x 106 cells/L
    2. Platelets greater than or equal to 100 x 109 cells/L
    3. Hemoglobin greater than or equal to 9 g/L.
11. Have the following chemistry levels at Baseline:

    1. AST (SGOT), ALT (SGPT) less than or equal to 1.5 x ULN
    2. Total bilirubin less than or equal to 1.5 ULN
    3. Creatinine less than or equal to 1.5 ULN; or 24-hour creatinine clearance greater than 60 mL/min
    4. Normal serum electrolytes and magnesium levels
12. Have a life expectancy of greater than or equal to 12 weeks.
13. Have an Eastern Cooperative Oncology Group (ECOG) Performance status of 0-2.
14. Patient or legal representative must understand the investigational nature of this study and sign an Independent Ethics Committee (EC)/Institutional Review Board (IRB)-approved written informed consent form (ICF) prior to receiving any study related procedure.

Exclusion Criteria:

1. Patient has radiographic evidence of active (symptomatic, untreated) intraparenchymal brain metastases; any meningeal metastases; or asymptomatic untreated intraparenchymal brain metastases requiring treatment.
2. Patient has received prior chemotherapy for metastatic prostate cancer.
3. Patient has a known infection with human immunodeficiency virus or active viral hepatitis.
4. Patient has active heart disease including myocardial infarction or congestive heart failure within the previous 6 months, symptomatic coronary artery disease, or uncontrolled arrhythmias.
5. Any condition which in the Investigator's opinion deems the patient an unsuitable candidate to receive study drug (e.g., uncontrolled bleeding or bleeding diathesis).
6. Any active infection requiring parenteral or oral antibiotics.
7. Patient treated with any of the following:

   1. Taxol, Taxotere or Abraxane for prostate cancer or any prior malignancy
   2. Concurrent radiation therapy (except for palliative radiotherapy for symptomatic bone metastasis which can be administered as clinically indicated)
8. Patient has pre-existing peripheral neuropathy of Grade greater than 1 based on the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-06; Primary Completion 2011-09 (Estimated); Study Completion 2011-09 (Estimated)

PRIMARY OUTCOMES:
Assessment of serum PSA | 1 year
  Measure serum PSA after 2, 4 and 6 cycles of treatment

SECONDARY OUTCOMES:
RECIST method assessment | 1 year
  Measurable soft tissue disease response based on the RECIST method, PFS, and OS will also be assessed after 2, 4 and 6 cycle to determine the treatment effectiveness with LE-DT after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Nancy A Dawson, M.D., Principal Investigator — Georgetown University; Brendan D Curti, M.D., Principal Investigator — Providence Health & Services
Locations (2):
- United States (2):
  - Georgetown University Medical center, Washington D.C., District of Columbia
  - Providence Portland Medical center, Portland, Oregon